CLINICAL TRIAL: NCT05045339
Title: Effectiveness of Ball Exercises on the Stereotypic Behavior of Children With Autism Spectrum Disorder
Brief Title: Ball Exercises and Stereotypic Behavior in Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Faisalabad (Other)
Responsible Party: Principal Investigator, Dr Izza Ayub; PT, Principal Investigator, University of Faisalabad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TUF/DR/DPT/157
Record Dates: First submitted 2021-09-06; First posted 2021-09-16 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Autism Spectrum Disorder
Keywords: ball exercises; physical therapy
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise Group (Experimental): Five different ball exercises were implemented for 35 minutes, 3 sessions per week for 2 months.
  Interventions: Procedure: Ball Exercises
- Control Group (No Intervention): No exercises were performed in control group

INTERVENTIONS:
Procedure: Ball Exercises — Different ball exercises which include stability ball roll, stability ball hug, catching, throwing was performed. Along with these exercises, ball tapping exercise was also performed.
  Arms: Exercise Group

SUMMARY:
Autism spectrum disorder (ASD) is a neuro-behavioral disorder associated with repetitive movements. The role of physical therapist towards an autistic child is most neglected one. Therefore, the objective of this study was to see the effectiveness of different ball exercise on stereotypic behavior of children with ASD. Different ball exercises were implemented for 2 months, 3 sessions per week and every session consist of 35 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed with ASD through experts
* Having recognized stereotypic behavior
* Having Intellectual Deficit (ID) and Attention Deficit Hyperactive Disorder (ADHD)
* Age ranging between 4-16 years
* Consented to take part

Exclusion Criteria:

* Having co-morbidities like schizophrenia and developmental delays
* Severe cases of ASD
* Showing aggressive behavior
* Having disease of cardiovascular or respiratory system
* Children unable to follow the command for exercise completely

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2025-02-09 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-05-28 (Actual)

PRIMARY OUTCOMES:
Stereotypic Behaviors | Two months
  Stereotypic behavior was the sole parameter assessed in this study using the Repetitive Behavior Scale-Revised (RBS-R), a well-established instrument known for its strong reliability and validity. The RBS-R was employed to evaluate self-stimulatory behaviors in children with Autism Spectrum Disorder (ASD). This 43-item questionnaire is organized into six distinct subscales, each targeting a specific dimension of repetitive behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Sidra Majeed; PT, Study Director — The University of Faisalabad
Locations (1):
- The University of Faisalabad, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No